CLINICAL TRIAL: NCT06087783
Title: PROtein, Leucine and Vitamin D Supplementation In Patients With GYnecologic Cancer Receiving First-line Platinum-based Chemotherapy
Brief Title: PROtein, Leucine and Vitamin D Supplementation In Patients With GYnecologic Cancer Receiving Platinum-based Chemotherapy
Acronym: PRODIGY-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Emanuele Cereda, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0014137/23
Record Dates: First submitted 2023-09-29; First posted 2023-10-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Gynecologic Cancer
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Single-group intervention study compared to matched historical controls
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Muscle-targeted nutritional support (Experimental): Two servings (40 grams each) of powder (Fortifit; Nutricia) which has to be dissolved in 125 ml of water. Per serving, 20 g whey protein, 3 g total leucine, 9 g carbohydrates, 3 g fat, 800 IU vitamin D, and a mixture of vitamins, minerals, and fibers.
  Interventions: Dietary Supplement: Experimental product - Fortifit® Powder
- Standard of care (Other): Control group receiving no nutritional intervention or on-demand non muscle-targeted nutritional intervention such as nutritional counseling with or without oral nutritional supplement
  Interventions: Other: Standard of care

INTERVENTIONS:
Dietary Supplement: Experimental product - Fortifit® Powder — Two servings (40 grams each) of powder (Fortifit®; Nutricia) which has to be dissolved in 125 ml of water. Per serving, 20 g whey protein, 3 g total leucine, 9 g carbohydrates, 3 g fat, 800 IU vitamin D, and a mixture of vitamins, minerals, and fibers.
  Other Names: Muscle-targeted nutritional support
  Arms: Muscle-targeted nutritional support
Other: Standard of care — Control group receiving no nutritional intervention or on-demand non muscle-targeted intervention such as nutritional counseling with or without oral nutritional supplement
  Arms: Standard of care

SUMMARY:
Open clinical trial addressing the effect of a nutritional support based on whey proteins, leucine and vitamin D on muscle mass and multiple anticancer treatment-related endpoints in patients with gynecologic cancer receiving first-line platinum-based chemotherapy (adjuvant or curative). A comparison to matched historical controls will be performed to address potential evidence of efficacy to be investigated in a subsequent randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of gynecologic cancer (ovarian, uterine, cervical);
* indication for a first-line chemotherapy (adjuvant or curative) with a platinum-based regimen to be used by investigator's choice within the framework of good clinical practice and in agreement with current Italian Association of Medical Oncology guidelines;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
* signed informed consent.

Exclusion Criteria:

* age <18 years
* ECOG performance status >2
* indication to or ongoing artificial nutrition support
* known kidney failure (previous glomerular filtration rate <30 ml/min);
* known liver failure (Child B or C)
* endocrine disorders associated with disorders of calcium metabolism (excluding osteoporosis)
* decompensated diabetes
* indications related to the study product: more than 10 µg (400 IU) of daily Vitamin D intake from medical sources More than 500 mg of daily calcium intake from medical sources; adherence to a high energy or high protein diet up or use of protein containing or amino acid containing nutritional supplements up to three months before starting the study.
* known allergy to milk, milk products or other components of the proposed interventions
* inclusion in other nutritional intervention trials
* patients refusal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Disease setting is gender-specific
Enrollment: 50 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in muscle mass area | 18 weeks
  Change in muscle mass at the end of first-line platinum-based chemotherapy (adjuvant or curative) evaluated with computed tomography scan at the level of the third lumbar vertebra

SECONDARY OUTCOMES:
Skeletal muscle mass | 18 weeks
  Change in skeletal muscle mass during the study evaluated with bioimpedance vectorial analysis
Body weight | 18 weeks
  Change in body weight during the study (assessed at each chemotherapy cycle)
Protein-calorie intake | 18 weeks
  Change in protein-calorie intake during the study (assessed at each chemotherapy cycle)
Handgrip strength | 18 weeks
  Change in handgrip strength
Treatment-related moderate-severe adverse events as assessed by Common Terminology Criteria for Adverse Events [CTCAE v5.0] | 18 weeks
  Difference in the incidence of grade >=3 toxicity, according to CTCAE v5.0. Toxicity is graded on 0-5 ordinal scale where a higher score means a worse outcome.
Adherence to treatment schedule | 18 weeks
  Difference in the proportion of patients completing the treatment schedule as planned
Total dose of chemotherapy administered | 18 weeks
  To be calculated as the percentage of chemotherapy dose administered with respect to the treatment plan
Patients requiring unplanned hospitalization | 18 weeks
  The rate of patients requiring unplanned hospitalization (one or more) during the study will be calculated
Tolerance to nutritional support | 18 weeks
  Occurrence of events of gastrointestinal intolerance

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Cereda, MD, PhD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- IRCCS San Matteo, Pavia, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided